CLINICAL TRIAL: NCT04566133
Title: Phase II Study of Combination of Trametinib (MEK Inhibitor) and Hydroxychloroquine (HCQ) (Autophagy Inhibitor) in Patients With KRAS Mutation Refractory Bile Tract Carcinoma (BTC).
Brief Title: Combination of Trametinib (MEK Inhibitor) and Hydroxychloroquine (HCQ) (Autophagy Inhibitor) in Patients With KRAS Mutation Refractory Bile Tract Carcinoma (BTC).
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tim Greten, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200152; 20-C-0152
Record Dates: First submitted 2020-09-25; First posted 2020-09-28 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Bile Duct Cancer; Biliary Cancer; Biliary Tract Neoplasms; Cholangiocarcinoma
Keywords: Tumor Regression; Progression Free Survival; New Drug Combination
MeSH Terms: conditions — Bile Duct Neoplasms; Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — trametinib; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort 1/Arm 1: Trametinib + Hydroxychloroquine (HCQ) (Experimental): Trametinib + hydroxychloroquine (HCQ)
  Interventions: Drug: Trametinib; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Trametinib — orally 2 mg once a day
  Other Names: Mekinist
Drug: Hydroxychloroquine — orally 600 mg twice a day-1,200 mg total dose
  Other Names: Plaquenil

SUMMARY:
Background:

Bile duct cancer is cancer of the slender tubes of the biliary tract. These tubes carry bile through the liver. Such cancer tumors often have an abnormal or mutated gene. Researchers think a mix of drugs can slow the progression of gene-mutated cancers of the biliary tract.

Objective:

To see if using a combination of trametinib and hydroxychloroquine (HCQ) increases the period of time it takes for a person s bile tract carcinoma (BTC) to get worse.

Eligibility:

Adults age 18 and older with BTC.

Design:

Participants will be screened with a physical exam, medical history, and cancer history. Their ability to do their normal activities will be assessed. They will have blood and urine tests. They will give a tumor sample. They will have heart tests. They may talk with a heart doctor. They may have an eye exam. They may have a tuberculosis test. They will have computer tomography (CT) scans of the chest, abdomen, and pelvis. They may have magnetic resonance imaging (MRI) scans of the chest, abdomen, pelvis.

Participants will repeat some screening tests throughout the study.

Participants will take HCQ and trametinib tablets by mouth daily in 28-day cycles. They will have study visits once a month. They will take the drugs until they have bad side effects or the drugs stop working.

Participants will have one more tumor biopsy during the treatment. They will have blood taken often.

One month after treatment ends, participants will have a safety follow-up visit. Then they will be called or emailed every 6 months for the rest of their life....

DETAILED DESCRIPTION:
Background:

* Among the new cases of bile tract carcinoma (BTC) that are diagnosed every year in the United States, there are approximately 6,500 cases of gallbladder carcinoma, 3,000 cases of extrahepatic cholangiocarcinoma, and 3,000 cases of intrahepatic cholangiocarcinoma.
* Current treatment options for patients with cholangiocarcinoma are limited and take no account of the known biological and genetic heterogeneity in these diseases. Median survival for advanced disease remains poor at approximately 1 year.
* Activating kirsten rat sarcoma (KRAS) mutations are frequently detected in all subtypes of BTC and can be found in up to 40% of BTC, predominantly in perihilar and distal cholangiocarcinoma (CCA). However, pharmacological inhibition of mutated KRAS has demonstrated little clinical benefit in general.
* Trametinib is a reversible, highly selective allosteric inhibitor of mitogen-activated extracellular signal regulated kinases methyl ethyl ketone 1 (MEK1) and methyl ethyl ketone 2 (MEK2). Tumor cells with KRAS mutations commonly have hyperactivated extracellular signal-related kinase (ERK) pathways in which activated MEK is a critical component. However, tumors are able to overcome MEK signaling inhibition by trametinib through upregulation of autophagy pathway.
* Hydroxychloroquine (HCQ) inhibits lysosomal acidification and prevents the degradation of autophagosomes, to suppress autophagy.
* Trametinib has been approved by FDA for the treatment of melanoma as a single agent or for the treatment of other cancers if tumors carry BRAF mutation. Hydroxychloroquine is approved for the treatment of malaria, lupus erythematosus and acute or chronic rheumatoid arthritis.
* Preclinical studies have shown that combined treatment of trametinib plus HCQ elicited striking tumor regression in animal model.

Objective:

-To determine whether the 5-month progression free survival (PFS) of the trametinib plus hydroxychloroquine (HCQ) combination in subjects with refractory bile tract carcinoma (BTC) with KRAS mutation exceeds 25%.

Eligibility:

* Histopathological confirmation of BTC or carcinoma highly suggestive of a diagnosis of BTC.
* Tumor must have KRAS mutation.
* Patients must have disease that is not amenable to potentially curative resection, transplantation or ablation.
* Age greater than or equal to 18 years
* Patients must have measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* At least two weeks washout period from previous therapy
* Eastern Cooperative Oncology Group (ECOG) less than or equal to 2
* Adequate renal, hepatic and bone marrow function

Design:

-The study is open-labeled phase 2 study. It is designed to enroll total 30 patients with refractory BTC, to test the hypothesis that treatment with a combination of HCQ and trametinib prevents cancer progression/recurrence. We propose that this combination will have relative safety profile and antitumor efficacy in BTC patients with KRAS mutation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histopathological confirmation of

  * biliary tract carcinoma (BTC) OR carcinoma in the setting of clinical and radiological characteristics which, together with the pathology, are highly suggestive of a diagnosis of BTC

Note: The term BTC includes intra- or extra- hepatic cholangiocarcinoma (CCA), gallbladder cancer or ampullary cancer.

* The tumor must have Kirsten rat sarcoma (KRAS) mutation(s) of clinical significance, confirmed by National Cancer Institute (NCI) Laboratory of Pathology or by Food and Drug Administration (FDA).
* Patients must have received or been intolerant of at least one line of chemotherapy.
* Patients must have at least 1 measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Patients must have disease that is not amenable to potentially curative resection, ablation or transplantation.
* Age greater than or equal to 18 years.
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-2
* If liver cirrhosis is present, patient must have a Child-Pugh score <7 (Class A)
* Patients must have adequate organ and marrow function as defined below:

  * absolute neutrophil count (ANC) greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * hemoglobin greater than or equal to 9 g/dL
  * total bilirubin if cirrhosis present: Part of Child Pugh requirement. If no cirrhosis: bilirubin should be less than or equal to 1.5 x upper limit of normal (ULN)
  * alanine aminotransferase (ALT) or aspartate aminotransferase (AST) less than or equal to 5 x ULN.
  * Creatinine OR Measured or calculated creatinine clearance (CrCl) (eGFR may also be used in place of CrCl)*** : < 1.5x institution upper limit of normal OR greater than or equal to 30 mL/min/1.73 m^2 for participant with creatinine levels greater than or equal to 1.5 X institutional ULN

Notes:

ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase);

AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase);

GFR=glomerular filtration rate; ULN=upper limit of normal.

***Creatinine clearance (CrCl) or estimated glomerular filtration rate (eGFR) should be calculated per institutional standard.

* Patients must have at least 1 focus of disease that is amenable to mandatory tumor biopsies and be willing to undergo this. Ideally, the biopsied lesion should not be one of the target measurable lesions, although this can be up to the discretion of the investigators.
* The study drugs are harmful for developing human fetus. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) at the study entry, for the duration of study treatment and up to 4 months after the last dose of the study drug(s). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Patients must be able to understand and be willing to sign a written informed consent.

EXCLUSION CRITERIA:

* Patients who have had standard-of-care anti-cancer therapy within 2 weeks of treatment initiation or therapy with investigational agents (e.g., chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies or other investigation agents), large field radiotherapy, or major surgery within 4 weeks of treatment initiation.
* Any unresolved toxicity NCI Common Terminology Criteria for Adverse Events (CTCAE) v.5 Grade greater than or equal to 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria. Patients with Grade greater than or equal to 2 neuropathy will be evaluated on a case-by-case basis.
* Has biliary duct obstruction, unless a treatable, clinically relevant obstruction has been relieved by internal endoscopic drainage/stenting, palliative by-pass surgery or percutaneous drainage prior to treatment initiation.
* Patients with known brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients with signs of liver failure, e.g., clinically significant ascites, encephalopathy, or variceal bleeding within six months before treatment initiation.
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyper viscosity or hypercoagulability syndromes)
* Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders: Congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias, stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 3 months before treatment initiation
  * History of glucose-6-phosphate dehydrogenase (G6PD) deficiency
  * History of seizures
  * Patients who are planning on embarking on a new strenuous exercise regimen after first dose of study treatment. Muscular activities, such as strenuous exercise, that can result in significant increases in plasma creatine kinase (CK) levels should be avoided while on study treatment
  * Patients who have neuromuscular disorders that are associated with elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
  * Impairment of gastrointestinal function or gastrointestinal disease (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection that under the judgment of the principal investigator (PI) may impair absorption of study drugs)
  * Any other condition that would, in the Investigator s judgment, contraindicate the patient s participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication (patients may not receive drug through a feeding tube), social/psychological issues, etc.
* Screening corrected QT interval by Fridericia's (QTcF) > 500 msec
* Known infection with human immunodeficiency virus (HIV), unless patient is on effective anti-retroviral therapy with undetectable viral load within 6 months of treatment initiation
* Known chronic hepatitis B virus, unless hepatitis B virus (HBV) viral load is undetectable.
* Known history of hepatitis C virus (HCV) infection, unless completed treatment and cured with undetectable HCV viral load.
* Known prior severe hypersensitivity to study drugs or any component in its formulations (CTCAE v5.0 grade >= 3).
* Pregnant women are excluded from this study because study therapy can cause fetal harm. Because there is potential risk for adverse events in nursing infants secondary to treatment of the mother with study therapy, breastfeeding should be discontinued if the mother is treated with study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing Plan (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0152.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1/Arm 1: Trametinib + Hydroxychloroquine (HCQ): Participants with bile tract carcinoma (BTC) or carcinoma in the setting of clinical and radiological characteristics which, together with the pathology, are highly suggestive of a diagnosis of BTC. Participants receive 2 mg of Trametinib orally once a day of every cycle, and 600 mg of hydroxychloroquine orally twice a day every cycle (1200 mg total dose).
Period: Overall Study
Arm/Group | Cohort 1/Arm 1: Trametinib + Hydroxychloroquine (HCQ)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cohort 1/Arm 1: Trametinib + Hydroxychloroquine (HCQ)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 41.95 (16.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: Participants with refractory bile tract carcinoma (BTC) with KRAS mutation that exceed 25% who receive trametinib plus hydroxychloroquine (HCQ) combination who are able to not have progressive disease at 5 months will be reported along with a 95% confidence interval. Progression was evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progression).
Time Frame: 3 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1/Arm 1: Trametinib + Hydroxychloroquine (HCQ)
Number analyzed (Participants) | 2
Months | 2.48 [NA to NA] — It is mathematically not possible to provide a confidence interval for 2 participants.

2. Secondary Outcome: Proportion of Participants With a Response (Complete Response (CR) + Partial Response (PR) Reported With an 80% Confidence Interval
Description: Response is defined as a Complete Response (CR) + Partial Response (PR) in participants with refractory BTC with KRAS mutation treated with the combination of trametinib plus HCQ. Response was evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete Response (CR) is disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. Any pathological lymph nodes must have reduction in short axis to <10 mm. Partial Response (PR) is at least a 30% decrease in the sum of target lesions, taking as reference the baseline sum diameters.
Time Frame: Every 2 months up to approximately 10 months
Measure: Number (80% Confidence Interval); unit: Proportion of participants
Arm/Group | Cohort 1/Arm 1: Trametinib + Hydroxychloroquine (HCQ)
Number analyzed (Participants) | 2
Proportion of participants
  Complete Response | 0 [0 to 0]
  Partial Response | 0 [0 to 0]

3. Secondary Outcome: Proportion of Participants With a Response (Complete Response (CR) + Partial Response (PR) Reported With an 95% Confidence Interval
Description: as for outcome 2
Time Frame: Every 2 months up to approximately 10 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1/Arm 1: Trametinib + Hydroxychloroquine (HCQ)
Number analyzed (Participants) | 2
proportion of participants
  Complete Response | 0 [0 to 0]
  Partial Response | 0 [0 to 0]

4. Secondary Outcome: Serious Adverse Events Possibly, Probably, and/or Definitely Related to Treatment
Description: Adverse events were assessed by the by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 90 days after treatment
Measure: Number; unit: adverse events
Arm/Group | Cohort 1/Arm 1: Trametinib + Hydroxychloroquine (HCQ)
Number analyzed (Participants) | 2
adverse events | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from start of treatment to death from any cause.
Time Frame: duration of time from the start of treatment to death from any cause, approximately 10 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1/Arm 1: Trametinib + Hydroxychloroquine (HCQ)
Number analyzed (Participants) | 2
Months | 3.1 [NA to NA] — It is mathematically not possible to provide a confidence interval for 2 participants.

6. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, assessed for approximately 3 months and 25 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1/Arm 1: Trametinib + Hydroxychloroquine (HCQ)
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events assessed from the date treatment consent signed to date off study, approximately 3 months and 25 days. Adverse Events monitored/assessed for approximately 3 months and 25 days; All-Cause Mortality monitored/assessed up to 10 months.
Description: The participants died due to their underlying disease.
Arm/Group | Cohort 1/Arm 1: Trametinib + Hydroxychloroquine (HCQ)
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1/Arm 1: Trametinib + Hydroxychloroquine (HCQ) (N=2)
Belching (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (4)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 1 (1)
Eosinophilia (Investigations) | 1 (2)
Lymphocyte count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, Two small pustule mouth lesions (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT04566133/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT04566133/ICF_001.pdf